CLINICAL TRIAL: NCT03360578
Title: Measuring Physiology in Individuals With Panic Disorder to Determine if Panic Attack Detection is Possible
Brief Title: Measuring Physiology to Determine if Pre-panic Attack Detection is Possible
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Psychology Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pre-Panic Physiology
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Garmin — A commercial grade health wearable

SUMMARY:
Participants will be asked to wear a physiological monitoring device for 1 week and record when panic events occur. Once the device is returned, the data will be downloaded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Panic disorder as described in the Diagnostic and Statistical Manual - 5 (DSM-5)

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18-65 individuals with panic disorder that are mentally capable to consent and are not pregnant
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Panic event | 1 year
  A timestamp of when a panic attack occurred
Heart Rate | 1 year
  Beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Psychology Center, Beverly, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided